CLINICAL TRIAL: NCT00361829
Title: Specificity of Mother-Infant Interaction: The Influence of Maternal Age, Employment Status, and Parenthood Status
Brief Title: The Influence of Maternal Age, Employment Status, and Parenthood Status on Children's Cognitive Development
Status: Completed | Type: Observational
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 880032; 88-CH-0032
Record Dates: First submitted 2006-08-08; First posted 2006-08-09 (Estimated); Last update posted 2026-01-15 (Actual); Status verified 2026-01-13

CONDITIONS: Child Development
Keywords: Childhood Growth and Development; Natural History

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Ecologic/Community: Married women, infants, caregivers, Japanese-American, Argentine-American

SUMMARY:
Research and theory tend to agree when suggesting that certain activities done by mothers have both immediate and delayed consequences for children's mental development in the first years of life.

The everyday interaction between an infant and a caregiver can be broken down into many categories. There are data linking both of these types of interaction to the mental development of children.

The study will focus on the extent to which maternal characteristics (age, employment status, parenthood status, and birth order of the child) influence the relation between maternal social and didactic caregiving and the social and mental development of children.

Mother-infant interaction will be observed when the infants are 5 months old.

When the children are 20 months old, measures of toddler function (e.g., ability to play and language development) and maternal behavior (e.g., encouragement of attention to the environment and I.Q.) will be obtained.

When the children are 48 months old, researchers will measure preschooler psychosocial functioning (e.g., I.Q., cognitive and social competencies) and maternal behavior (e.g., "scaffolding").

Understanding the relation between children's experiences as infants, toddlers, and preschoolers and their eventual intellectual and social functioning is an essential part of normal developmental research.<TAB>

DETAILED DESCRIPTION:
Research and theory concur in suggesting that certain maternal activities have both immediate and protracted consequences for children's cognitive development in the first years of life. Two conceptually distinct categories of caretaker-child interactions can be identified: social and didactic. These encompass much of the everyday behavior of infants' caretakers. There are data linking both of these types of behavior to cognitive development in children. In previous work we have investigated these relations in early infancy using samples of convenience. In the proposed study set, this work will be replicated and extended by focusing on the extent to which the characteristics of maternal age, employment status, parenthood status and birthorder of the child influence observed relations between maternal, social and didactic caretaking on the one hand and infant, toddler, preschool age, and middle childhood, and adolescent social and cognitive competencies on the other. For a subset of infants of employed mothers, their substitute caregivers will be added to the sample. Understanding the full range of experience for those infants with multiple caregivers is important in the context of a study designed to elucidate dimensions of experience that influence social and cognitive development. Naturalistic mother-infant interaction will be observed when infants are 5 months old. When study participants are 20 months old, measures of toddler functioning (e.g., play competence and language development) and maternal behavior (e.g., encouragement of attention to the environment, I.Q.) will be obtained. At 48 months, measures of preschooler psychosocial functioning (e.g., I.Q., cognitive and social competencies) and maternal behavior (e.g., "scaffolding") will be obtained. At age 10 and 14 years, data assessing the child's adjustment, development, and functioning in multiple areas will be obtained from the child, both parents, and the schoolteacher (age 10 only). Measures of parental attitudes and family functioning will also be obtained. Theoretical formulations about how specific parent-child interactions may contribute to cognition have challenged investigators to look beyond demographic variables as markers of parental stimulation and to consider specific relations between types of interactions and the acquisition of particular skills at different points in time. Understanding the mechanisms linking experience in early infancy through toddlerhood, the preschool years, middle childhood and early adolescence with intellectual and social functioning is an essential aspect of normative developmental research. In addition, examining these phenomena cross-culturally will contribute importantly to our understanding of children and their families.

ELIGIBILITY:
* INCLUSION CRITERIA:

All subjects are normal volunteers.

At initial recruitment, all mothers will be married women living in intact families with healthy, full-term, first-born infants. Most will be living in intact families.

Prior to inclusion in the sample, basic demographic information will be obtained for all study participants including substitute caregivers but excluding school teachers. Variables include age, race, cultural background, primary language, marital status, SES (as assessed by the Hollingshead Four-Factor Index of Social Status, 1975), and educational level. In addition, for caregivers, information about their experience caring for children and about the peer environment, including the number of children routinely present, their sexes, and their ages, will be obtained.

To the extent that the adolescent sample diverges from sample criteria with respect to marital status and SES, appropriate controls will be used.

Subjects in the Argentine-American and Japanese-American project will be selected to represent families high vs low on appropriate measures of acculturation.

The healthy second born infants of 80 mothers already enrolled in the protocol will also be recruited into the sample at the time of their birth. These infants will be selected to comprise four equal groups based on the gender composition of the sibling dyad: male/male, male/female, female/female, and female/male.

Ages: 5 Months to 23 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Mother-infant interaction will be observed when the infants are 5 months old. When the children are 20 months old, measures of toddler function (e.g., ability to play and language development) and maternal behavior (e.g., encouragement of attention to the environment and I.Q.) will be obtained. When the children are 48 months old, researchers will measure preschooler psychosocial functioning (e.g., I.Q., cognitive and social competencies) and maternal behavior (e.g., "scaffolding").
Sampling Method: Non-Probability Sample
Enrollment: 2355 (Actual)
Dates: Start 1988-02-17 (Actual)

PRIMARY OUTCOMES:
Measures of child adaptive functioning | 5, 20,and 48 months, 10 years, 14 years, 18 years, and 23 years
  Measures of child adaptive functioning

CONTACTS AND LOCATIONS:
Overall Officials: Diane L Putnick, Ph.D., Principal Investigator — Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD)
Locations (4):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States
- Federal University of Rio de Janeiro-Participants Homes, Rio de Janeiro, Brazil
- University of Bamenda, Cameroon-Participants Homes, Bamenda, Cameroon
- University of Saskatchewan-Participants Homes, Saskatchewan, Canada

IPD SHARING:
Plan to Share IPD: No
The protocol does not make mention of IPD sharing.

REFERENCES:
- [Background] Rowe A. Characteristics of hospital care. Nurs Times. 1969 Oct 23;65(43):1376-7. No abstract available. PMID 5823787
- [Background] Kuiumdzhieva A, Denchev D. [ATP yield from yeasts of the genera Candida and Torulopsis cultured in a chemostat on a methanol medium]. Acta Microbiol Bulg. 1984;15:50-5. No abstract available. Bulgarian. PMID 6541423
- [Background] Smith WL, Egle JL Jr, Adams MD. Adrenergic receptors in the nucleus tractus solitarii of the rat. Eur J Pharmacol. 1982 Jun 16;81(1):11-9. doi: 10.1016/0014-2999(82)90596-9. PMID 6126366
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_1988-CH-0032.html